CLINICAL TRIAL: NCT03354455
Title: Targeting the Pre-supplementary Motor Area With Repetitive Transcranial Magnetic Stimulation to Alleviate Levodopa-induced Dyskinesia in Parkinson´s Disease
Brief Title: Investigating the Causal Role of preSMA in Levodopa-induced Dyskinesia in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Danish Movement Disorder Society (DANMODIS) (Unknown); Danish Parkinson Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-15017863
Record Dates: First submitted 2017-06-01; First posted 2017-11-28 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-08

CONDITIONS: Dyskinesia, Drug-Induced; Parkinson Disease
MeSH Terms: conditions — Dyskinesia, Drug-Induced; Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sham stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REAL TMS (Experimental): 30 minutes of repetitive transcranial magnetic stimulation with 100% of the patients' individual resting motor threshold.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- SHAM TMS (Sham Comparator): 30 minutes of repetitive transcranial magnetic stimulation with 30% of the patients' individual resting motor threshold.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Frequency: 1 Hz., Pulse shape: biphasic, Duration: 30 minutes (1800 pulses).
  Neuronavigation: MRI-guided and robot-assisted neuronavigation using Localite software and an Axilum robot.

SUMMARY:
Using a within-subject cross-over design, we will include 20 patients with Parkinson disease (PD) and peak-of-dose dyskinesia.

Patients will be studied after withdrawal from their normal dopaminergic medication.

On two separate days, each patient will receive off-line, effective (high-intensity) or ineffective (low-intensity) 1 Hz repetitive transcranial magnetic stimulation (rTMS) of the presupplementary motor area (preSMA) before functional magnetic resonance (fMRI). Immediately after the patient will perform a Go/No-Go task during fMRI in the the OFF state for 9 minutes. Then the scan is paused and the patient will receive 200 mg fast-acting oral levodopa and undergo whole-brain task-related fMRI at 3 Tesla until peak-of-dose dyskinesia will emerge.

During task-related fMRI, patients has to click on a mouse with their right hand (Right-Go), left hand (Left-Go), or no action (No-Go) in response to arbitrary visual cues.

The patients will also be tested for different aspects of impulsivity using neuropsychological questionnaires and computerized tests.

DETAILED DESCRIPTION:
The most common form of levodopa-induced dyskinesias (LID) manifests when levodopa levels are highest and is referred to as peak-of-dose dyskinesia. 50% of patients experience LID after 4-6 years of treatment, reaching a frequency of 40% after 4-6 years. The main risk factors for developing LID are disease duration, levodopa dose and age-at-onset, but none of these factors alone can predict whether and when an individual patient with PD will develop LID. There is converging evidence that exogenously administered levodopa induces non-physiological release and reuptake of dopamine in the striatum. This non-physiological dopaminergic stimulation gives rise to aberrant plasticity in the striatum that causes a sensitization of the cortico-basal ganglia system to levodopa. Dyskinesia often severely affects patients' quality of life requiring advanced treatment.

Adopting a novel pharmacological fMRI (ph-fMRI) approach, our group recently identified a functional signature of LID in the human brain: To bypass any problems due to movement artefacts, fMRI was performed in the time-span between the administration of levodopa and the onset of dyskinesia. Ph-fMRI revealed that a single oral dose of levodopa caused an abnormal cortico-striatal activation and connectivity pattern in pre-SMA and putamen in LID patients relative to PD patients without LID. We predict that 1 Hz rTMS of pre-SMA will attenuate the levo-dopa-induced overactivity in the pre-SMA and putamen and normalise the pre-SMA-putamen connectivity pattern. This may possibly involve an altered interaction with the right inferior frontal gyrus (rIFG).On two separate days, each patient will receive effective (high-intensity) or ineffective (low-intensity) 1 Hz rTMS (i.e. control rTMS session) of the pre-SMA before fMRI (Off-line rTMS).

Pharmacological fMRI (ph-fMRI): Immediately after rTMS the patient will perform a Go/No-Go task during fMRI in the the OFF state for 9 minutes. Then the scan is paused and the patient will receive 200 mg fast-acting oral levodopa and undergo whole-brain task-related fMRI at 3 Tesla until peak-of-dose dyskinesia will emerge. During task-related fMRI, patients press a computer mouse with the right hand (Right-Go), left hand (Left-Go), or no action (No-Go) in response to arbitrary visual cues.

We want to include 20 patients in the final analysis of the study. In a previous comparable study we experienced a drop-out rate around a third. We therefore aim to enrol 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease (Hoehn & Yahr 1-3)
* Peak-of-dose levodopa-induced dyskinesia

Exclusion Criteria:

* Insufficient Danish language skills
* Neurological disease other than Parkinson's Disease
* Major psychiatric illness
* Sedatives or serotonergic medication in their current treatment.
* Severe tremor
* Montreal Cognitive Assessment score < 26

Contraindication for transcranial magnetic stimulation:

* Epilepsy or epilepsy in 1st degree relatives
* Contraindications for MRI-scanning:
* Pacemaker
* Pregnancy
* Metallic foreign objects inside the body
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-09-16 (Actual); Study Completion 2018-09-16 (Actual)

PRIMARY OUTCOMES:
Levodopa-induced change in task-related regional neural activity as indexed by the blood oxygen level dependent (BOLD) signal | Within the first 60 minutes after levodopa intake
  A single priming session of REAL rTMS over the preSMA will attenuate the abnormal pharmacodynamic BOLD response (which is an index of regional neural activity) in the cortico-basal ganglia loop after levodopa challenge compared with SHAM rTMS.

SECONDARY OUTCOMES:
Onset of LID | Within the first 60 minutes after levodopa intake
  A single priming session of REAL rTMS over the SMA will prolong the time to onset of LID compared with SHAM.
Severity of LID | Within the first 60 minutes after levodopa intake
  A single priming session of REAL rTMS over the SMA will lower the the severity of LID measured on the Unified Dyskinesia Rating Scale (UDysRS) compared with SHAM.

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig R Siebner, MD, DMSci, Principal Investigator — Danish Research Centre for Magnetic Resonance
Locations (1):
- Danish Research Centre for Magnetic Resonance, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided